CLINICAL TRIAL: NCT02426138
Title: Community Servings: Food as Medicine for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Seth A Berkowitz, Instructor in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014P002778
Record Dates: First submitted 2015-03-07; First posted 2015-04-24 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Med. Tailored Meal Delivery, Usual Care + Choose Myplate (Experimental): Participants will receive 12 weeks of medically tailored meal delivery, comprising approximately half of their weekly caloric intake and consisting of foods prepared under the supervision of a registered dietitian to be compatible with a diabetes diet. They will also receive usual diabetes care and a Choose MyPlate healthy eating brochure for 12 weeks.
  Interventions: Other: Medically Tailored Meal Delivery (MTM); Other: Usual Care + Choose MyPlate
- Usual Care + Choose Myplate, Med. Tailored Meal Delivery (Active Comparator): Participants will receive usual diabetes care and a Choose MyPlate healthy eating brochure for 12 weeks.
  Interventions: Other: Usual Care + Choose MyPlate

INTERVENTIONS:
Other: Medically Tailored Meal Delivery (MTM) — Patients will receive delivery of medically tailored meals for 12 weeks
  Arms: Med. Tailored Meal Delivery, Usual Care + Choose Myplate
Other: Usual Care + Choose MyPlate — Patients will receive usual diabetes care + a Choose MyPlate healthy eating brochure for 12 weeks

SUMMARY:
Food insecurity, defined as difficulty accessing food owing to cost, affects 1 in 5 diabetes patients. To address this, the investigators are conducting a pilot randomized controlled trial of medically tailored meal delivery (MTM). The pilot study has two specific aims:

Aim 1: To determine the effect of receiving MTM on dietary quality for food insecure diabetes patients with hyperglycemia Aim 2: To determine the feasibility and acceptability of the program as a medical intervention and refine the program as needed for testing in larger studies.

This study is a crossover randomized controlled pilot trial, where approximately 50 participants, 25 in each arm, will be randomized to receipt of 12 weeks of MTM, to begin immediately, or waitlist control. After 12 weeks, the groups will crossover, with the waitlist control group now receiving 12 weeks of MTM. At baseline, 12 weeks, and 24 weeks, the participants will complete assessments of their dietary quality (HEI score), psychosocial measures such as diabetes distress and food insecurity, along with measures of body mass index, blood pressure, hemoglobin A1c, and lipids.

DETAILED DESCRIPTION:
a. Historical background The Center for Disease Control and Prevention (CDC) estimates that there are currently 29 million people with diabetes and 86 million people with pre-diabetes in the U.S. One in 10 Americans has diabetes now, and, if current trends continue, 1 in 3 Americans will have diabetes by 2050. This chronic disease significantly impacts both quality of life and rapidly rising national healthcare costs. The estimated cost of diabetes in the U.S. in 2014 was $265 billion with $176 billion in direct medical costs and $89 billion is indirect medical costs (disability, work loss, premature mortality). Medical expenses for people with diabetes are 2.3 times higher than for people without diabetes.

Food insecurity, defined as limited access to nutritious food due to cost, has been associated with increased prevalence of diabetes and worse diabetes control. Food insecurity may worsen diabetes by decreasing consumption of fresh fruits and vegetables and increasing consumption of inexpensive, calorie-dense food, and which in turn leads to greater Hemoglobin A1c, an indicator of hyperglycemia, over time.

c. Rationale behind the proposed research, and potential benefits to participants and/or society

Approximately 20% of diabetes patients report food insecurity, a number that increases to over 25% among those with the worst metabolic control.5 The prevalence of food insecurity is also 20% in the MGH Population we surveyed (data not yet published). Hyperglycemia is particularly responsive to dietary changes,8 yet few interventions have attempted to address food insecurity in diabetes care. Prior studies have examined the impact of the Supplemental Nutrition Assistance Program (SNAP, formerly the Food Stamp Program), but have not found important improvements in diabetes outcomes for participants9. This may be because neighborhood access to produce and other high quality food is low for many SNAP participants, or because making healthy food choices is difficult in resource-constrained environments. Additionally, recent sociological work has shown that expecting low-income women to cook healthy meals for their families induces a significant burden, and the burden of these expectations may drive less healthy food choices. Additionally, while significant time is needed for healthy food preparation, low-income patients often face limited leisure time, and multiple competing demands for both time and financial resources. Alternatively, direct provision of healthy foods was incidentally noted to improve diabetes outcomes in a prior randomized controlled trial, but this study was not conducted with the goal of addressing food insecurity.

In this study, we propose to test whether home delivery of freshly prepared meals specifically tailored to the needs of diabetes patients improves their dietary quality. We hypothesize that the delivery of the meals will help them eat more healthily and improve the food security of participants. Secondary outcomes in this pilot study will be weight and metabolic control, along with psychological aspects of diabetes care.

Aim 1: To evaluate the effectiveness of receiving Community Servings meals on dietary quality for food insecure diabetes patients with severe hyperglycemia (HbA1c > 8.0%) H1. Primary outcome. Healthy Eating Index 2010 (HEI) score: We hypothesize that the CS group will demonstrate greater improvements in dietary quality, as assessed by HEI score, at 12 weeks, compared with usual care. The sample size of 50 provides 80% power to detect a 5 point difference between the CS and usual care groups, assuming an 11 point standard deviation and accounting for a 10% drop-out rate.

H1b. Secondary exploratory outcomes. Medical outcomes: We hypothesize that compared with usual care, CS group participants will improve HbA1c, blood pressure, weight, and lipids from baseline at the end of the intervention.

H1c. Behavioral and psychosocial outcomes: Because meal provision will reduce stress related to procuring healthy meals, and free up household resources that would otherwise be spent on food, we hypothesize that compared with usual care, the CS groups will have greater improvements from baseline in patient-reported outcomes of diabetes distress and material need security.

Aim 2: To evaluate the feasibility of providing meals and patient experience with the CS program, particularly focusing on factors that determine acceptability, continuation, and scalability We will use a mixed methods approach using participant structured interviews and surveys to assess engagement and satisfaction with the program, and participant interviews or focus groups to compare responders and non-responders. We will also collect quantitative indicators of feasibility and implementation such as percent of meals delivered and consumed, enrollment and persistence with the program, and logistical issues in order to plan for a future full-scale intervention.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of type 2 diabetes

  * Age 18 years or older
  * HbA1c level >8.0%
  * Report food insecurity as indicated by the 2-item USDA Food Security Survey Module13
  * Willing to commit to random assignment to either receive CS meals immediately or as a waitlist control
  * Stable health, with no severe medical comorbidities that might interfere with their ability to participate in the intervention, such as severe psychiatric illness or imminent hospitalization
  * Be willing to keep a food diary
  * Be willing to attend and complete a baseline, 12 week, and 24 week assessment at MGH
  * Be able to understand and communicate effectively in English
  * Have a primary care physician within the MGH practice based research network
  * Live in an area where Community Servings can deliver meals
  * Ability to store and prepare Community Servings meals

Exclusion Criteria:

* • Must not be pregnant or planning pregnancy in the next year

  * Currently enrolled in another diabetes study Food allergy that would prohibit consumption of meals
  * Receiving episodic treatments that may increase blood glucose levels (e.g. prednisone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth A Berkowitz, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berkowitz SA, Delahanty LM, Terranova J, Steiner B, Ruazol MP, Singh R, Shahid NN, Wexler DJ. Medically Tailored Meal Delivery for Diabetes Patients with Food Insecurity: a Randomized Cross-over Trial. J Gen Intern Med. 2019 Mar;34(3):396-404. doi: 10.1007/s11606-018-4716-z. Epub 2018 Nov 12. PMID 30421335
- [Derived] Berkowitz SA, Shahid NN, Terranova J, Steiner B, Ruazol MP, Singh R, Delahanty LM, Wexler DJ. "I was able to eat what I am supposed to eat"-- patient reflections on a medically-tailored meal intervention: a qualitative analysis. BMC Endocr Disord. 2020 Jan 20;20(1):10. doi: 10.1186/s12902-020-0491-z. PMID 31959176

RESULTS

PARTICIPANT FLOW:
Groups:
- Meal Delivery Then Usual Care + Choose myPlate: During the first intervention period, participants in this arm will receive 12 weeks of medically tailored meal delivery, comprising approximately half of their weekly caloric intake and consisting of foods prepared under the supervision of a registered dietitian to be compatible with a diabetes diet. They will also receive usual diabetes care and a Choose MyPlate healthy eating brochure. Data recorded during or at the end of the first intervention period will comprise the 'on-meal' data for this participants in this arm.
  Following this, during the second intervention period, they will receive 12 weeks of usual diabetes care + a Choose MyPlate healthy eating brochure, without meal delivery. Data recorded during or at the end of the second intervention period will comprise the 'off-meal' data for participants in this arm.
- Usual Care + Choose myPlate Then Meal Delivery: During the first intervention period, participants in this arm will receive 12 weeks of usual diabetes care + a Choose MyPlate healthy eating brochure, without meal delivery. Data recorded during or at the end of the first intervention period will comprise the 'off-meal' data for participants in this arm.
  Following this, during the second intervention period, participants will receive 12 weeks of medically tailored meal delivery, comprising approximately half of their weekly caloric intake and consisting of foods prepared under the supervision of a registered dietitian to be compatible with a diabetes diet. They will also receive usual diabetes care and a Choose MyPlate healthy eating brochure. Data recorded during or at the end of the second intervention period will comprise the 'on-meal' data for this participants in this arm.
Period: First Intervention (12 Weeks)
Arm/Group | Meal Delivery Then Usual Care + Choose myPlate | Usual Care + Choose myPlate Then Meal Delivery
Started | 21 | 23
Completed | 20 | 22
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention (12 Weeks)
Arm/Group | Meal Delivery Then Usual Care + Choose myPlate | Usual Care + Choose myPlate Then Meal Delivery
Started | 20 | 22
Completed | 20 | 22
Not Completed | 0 | 0
Period: Intent to Treat Population Milestone
Arm/Group | Meal Delivery Then Usual Care + Choose myPlate | Usual Care + Choose myPlate Then Meal Delivery
Started | 20 | 22
Completed | 20 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meal Delivery Then Usual Care + Choose myPlate | Usual Care + Choose myPlate Then Meal Delivery | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.66 (12.25) | 59.21 (13.11) | 58.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 10 | 13 | 23
  Non-Hispanic Black | 5 | 6 | 11
  Hispanic | 4 | 3 | 7
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42
Healthy Eating Index 2010 Score [Mean (Standard Deviation); unit: units on a scale] — Calculated using data from ASA24 24-hour dietary recall tool Healthy Eating Index 2010 Score Minimum and Maximum range = 0 to 100 Higher scores indicate better diet quality
  units on a scale | 57.27 (14.65) | 57.16 (13.49) | 57.21 (14.04)

OUTCOME MEASURES:

1. Primary Outcome: Healthy Eating Index 2010 Score
Description: Calculated using data from ASA24 24-hour dietary recall tool Healthy Eating Index 2010 Score Minimum and Maximum range = 0 to 100 Higher scores indicate better diet quality The score is an average of the three-time periods that data was collected
Time Frame: Average of 3 24-hour food recalls per study period (on and off meals; one in-person visit and 2 over the phone at 4 and 8 weeks into the study)
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- On Meals: Outcome recorded while receiving medically tailored meals
- Off Meals: Outcome recorded while not receiving meals
Arm/Group | On Meals | Off Meals
Number analyzed (Participants) | 31 | 39
units on a scale | 71.30 (7.49) | 39.89 (7.80)

2. Secondary Outcome: Number of Participants With Food Insecurity
Description: Food insecurity is defined as > 2 affirmative responses on the 10 adult referenced items USDA Household Food Security Survey Module
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- On-Meals: Outcome recorded while receiving medically tailored meals
- Off-Meals: Outcome recorded while not receiving meals
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 39
Participants | 13 | 24

3. Secondary Outcome: Diabetes Distress Scale
Description: Diabetes Distress calculated using the Diabetes Distress Scale Minimum and Maximum scores range of the scale is 17-106 For this measure the lower the score the better
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 34
units on a scale | 30.94 (13.77) | 30.82 (10.70)

4. Other Pre Specified Outcome: Hemoglobin A1c
Description: This will be measured using a fasting blood draw at baseline, 12 and 24 weeks
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: ITT
Measure: Mean (Standard Deviation); unit: % of hemoglobin
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 39
% of hemoglobin | 7.99 (1.86) | 8.15 (1.72)

5. Other Pre Specified Outcome: LDL Cholesterol
Description: A fasting blood draw will be used to measure: LDL Cholesterol
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: ITT
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 39
mg/dl | 97.54 (35.67) | 101.43 (43.11)

6. Other Pre Specified Outcome: Body Mass Index
Description: Body Mass Index will be measured in light street clothes (without shoes) using a single calibrated scale.
  Height measured using a stadiometer. Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters.
  A high BMI can be an indicator of high body fatness.
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: ITT
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 39
kg/m^2 | 34.24 (6.76) | 34.79 (6.97)

7. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Measured using a calibrated sphygmomanometer with appropriate cuff sizes based on arm circumference. Average of 2 readings, first manual and second automated at 1 min intervals following a 5 min period of rest.
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant using a calibrated sphygmomanometer
Population: ITT
Measure: Mean (Standard Deviation); unit: mm hg
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 39
mm hg | 133.04 (17.60) | 136.00 (18.77)

8. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: as for outcome 7
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant using a calibrated sphygmomanometer
Population: ITT
Measure: Mean (Standard Deviation); unit: mm hg
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 39
mm hg | 76.86 (8.65) | 78.16 (10.11)

9. Other Pre Specified Outcome: Change From Baseline in Medication Adherence
Description: Change from baseline in Medication Adherence Rating Scale (Assessed using medication adherence rating scale) Range is 0-25 The higher the number the better
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 39
units on a scale | 23.19 (2.86) | 22.28 (3.21)

10. Other Pre Specified Outcome: Number of Participants With Cost Related Medication Under-Use
Description: Cost Related Medication Under-use (Defined as > 0 affirmative responses to 4-items on cost-related medication under-use from the medication expenditure panel survey)
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 39
Participants | 7 | 11

11. Other Pre Specified Outcome: Number of Participants With Food and Medication Trade-offs
Description: Prevalence of food and medication trade-offs between groups
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 39
Participants | 9 | 9

12. Other Pre Specified Outcome: Depressive Symptoms (Assessed Using the PHQ-8 Scale)
Description: Patient Health Questionnaire - 8 item version. The score ranges 0-24, The lower score represents less depressive symptoms
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 31 | 39
units on a scale | 6.16 (5.15) | 6.13 (4.96)

13. Other Pre Specified Outcome: Change From Baseline in Cognitive Burden (Assessed Using Times on the Stroop Task)
Description: This outcome was planned to be measured but not measured owing to technical difficulties in assessment
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: This outcome was planned to be measured but not measured owing to technical difficulties in assessment
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Number of Participants With Self-reported Hypoglycemia
Description: Report of hypoglycemia requiring assistance in last 3 months
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | On-Meals | Off-Meals
Number analyzed (Participants) | 30 | 36
Participants | 14 | 23

15. Other Pre Specified Outcome: Triglycerides
Description: A fasting blood draw will be used to measure: Triglycerides
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant by fasting blood draw
Population: ITT
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | On Meals | Off Meals
Number analyzed (Participants) | 31 | 39
mg/dl | 142.00 [83.00 to 258.00] | 127.50 [99.5 to 175.5]

16. Other Pre Specified Outcome: HDL Cholesterol
Description: A fasting blood draw will be used to measure: HDL Cholesterol
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant by fasting blood draw
Population: ITT
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | On Meals | Off Meals
Number analyzed (Participants) | 31 | 39
mg/dl | 45.81 (11.23) | 46.36 (10.20)

17. Other Pre Specified Outcome: Total Cholesterol
Description: A fasting blood draw will be used to measure: Total Cholesterol
Time Frame: Measured at end of On-Meals Period and end of Off-Meals Period for each participant by fasting blood draw
Population: ITT
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | On Meals | Off Meals
Number analyzed (Participants) | 31 | 39
mg/dl | 182.63 (47.30) | 178.69 (43.82)

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Medically Tailored Meal Delivery: Participants will receive 12 weeks of medically tailored meal delivery, comprising approximately half of their weekly caloric intake and consisting of foods prepared under the supervision of a registered dietitian to be compatible with a diabetes diet. They will also receive usual diabetes care and a Choose MyPlate healthy eating brochure.
  Medically Tailored Meal Delivery (MTM): Patients will receive delivery of medically tailored meals for 12 weeks
  Usual Care + Choose MyPlate: Patients will receive usual diabetes care + a Choose MyPlate healthy eating brochure
- Usual Care + Choose Myplate (Delayed): Participants will receive usual diabetes care and a Choose MyPlate healthy eating brochure for 12 weeks.
  Usual Care + Choose MyPlate: Patients will receive usual diabetes care + a Choose MyPlate healthy eating brochure
  They will then receive 12 weeks of medically tailored meal delivery, comprising approximately half of their weekly caloric intake and consisting of foods prepared under the supervision of a registered dietitian to be compatible with a diabetes diet
Arm/Group | Medically Tailored Meal Delivery | Usual Care + Choose Myplate (Delayed)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

LIMITATIONS AND CAVEATS:
Short-term study designed to test change in diet quality only. Not designed for clinical endpoints Single center study in one region of US

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT02426138/Prot_SAP_000.pdf